CLINICAL TRIAL: NCT05723185
Title: Primary Care-Hospital Embedding: a Prospective, Multicentric, Observational Study
Acronym: PRIME
Status: Active, not recruiting | Type: Observational
Sponsor: Rovere Querini Patrizia (Other)
Collaborators: ASST Fatebenefratelli Sacco (Other); ASST Grande Ospedale Metropolitano Niguarda (Other)
Responsible Party: Sponsor-Investigator, Rovere Querini Patrizia, Director, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: PRIME
Record Dates: First submitted 2023-02-03; First posted 2023-02-10 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure; Chronic Obstructive Pulmonary Disease; Diabetes Mellitus; Pneumonia; Urinary Tract Infections; Fever of Unknown Origin; Deep Vein Thrombosis; Hypertension
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus; Pneumonia; Urinary Tract Infections; Fever of Unknown Origin; Venous Thrombosis; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Internal medicine model: This group of patients will be treated at the outpatient clinic which is run by internal medicine specialists
  Interventions: Other: Outpatient visit
- Specialist model: This group of patients will be treated at the outpatient clinic which is run by cardiologists and/or diabetologists
  Interventions: Other: Outpatient visit

INTERVENTIONS:
Other: Outpatient visit — Patients will be seen and treated at the outpatient clinic like in the usual care

SUMMARY:
This is a multicentric, prospective, observational study with two cohorts and adjunctive procedure. It aims at collecting and analyzing data about the function of an innovative hospital-territory integration health service for the management of patients with intermediate urgency, or emergency department "white codes." This service, activated in the participating centers, will be provided in two alternative modalities, one so-called "dual specialty" (cardiology and diabetes specialist outpatient clinic) and a second one more focused on the figure of the specialist in Internal Medicine.

The investigators will monitor the population treated in these centers (presenting complaint, medical history, clinical-radiological data, performed therapies and overall health path) and the degree of satisfaction of the General Practitioners who sent their patients there and the degree of satisfaction of the patients themselves. The data collected will also be used to evaluate the effectiveness of the outpatient clinics in terms of reducing improper admissions to the Emergency Departments and hospitalizations. The two modes of service delivery will be compared.

This is an 18-month study, sponsored by our Scientific Directorate and carried out on a nonprofit basis. The study will enroll 246 patients and 30 healthy volunteer General Practitioners. The clinical trial will be conducted in accordance with Good Clinical Practice standards.

ELIGIBILITY:
Inclusion Criteria:

* Patients sent by General Practitioners for outpatient evaluation in the two models
* Patients able to read and sign the informed consent
* Patients able to read and fill the questionnaire

Exclusion Criteria:

- Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated at the outpatient clinics (one cardio-diabetes specialty managed, one internist managed) with direct access for intermediate emergency management. For San Raffaele Hospital, patients will be those treated at the strategic project of hospital-territory embedding at Ville Turro (Milan). General practitioners (GPs) in the Milan Metropolitan Area will be recruited for questionnaire filling and patients referral.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Analyse and compare the function of the two outpatient clinic models | 6 months for each subject
  We will gather data describing the different patients treated at the two outpatient clinics; moreover, we will describe the timing, efficiency and effectiveness of the interventions and compare the two models; lastly, feedback from patients and general practitioners will be gathered through questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sundmacher L, Fischbach D, Schuettig W, Naumann C, Augustin U, Faisst C. Which hospitalisations are ambulatory care-sensitive, to what degree, and how could the rates be reduced? Results of a group consensus study in Germany. Health Policy. 2015 Nov;119(11):1415-23. doi: 10.1016/j.healthpol.2015.08.007. Epub 2015 Sep 2. PMID 26428441
- [Background] De Lorenzo R, Montagna M, Bossi E, Vitali G, Taino A, Cilla M, Pata G, Lazorova L, Pesenti R, Pomaranzi C, Bussolari C, Martinenghi S, Bordonaro N, Di Napoli D, Rizzardini G, Cogliati C, Morici N, Rovere-Querini P. A Pilot Study of the Efficacy and Economical Sustainability of Acute Coronavirus Disease 2019 Patient Management in an Outpatient Setting. Front Med (Lausanne). 2022 Apr 27;9:892962. doi: 10.3389/fmed.2022.892962. eCollection 2022. PMID 35572976
- [Background] Montagna M, Morici N, Tritschler T, Rovere Querini P. Fostering the intersection between primary care and hospital: hints from a survey and the PRIME (PRIMary care-hospital Embedding) project. Eur J Intern Med. 2023 Mar;109:131-134. doi: 10.1016/j.ejim.2022.10.023. Epub 2022 Nov 3. No abstract available. PMID 36334984